CLINICAL TRIAL: NCT05900349
Title: Carbohydrate Mouth Rinses and Caffeine Gum Increase the Romanian Deadlift Performance on the Flywheel Training Device: A Randomised, Cross-Over Study
Brief Title: Carbohydrate Rinsing and Caffeine Gum on Performance of Romanian Deadlifts Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 111-2
Record Dates: First submitted 2023-03-24; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Carbohydrate; Caffeine
Keywords: Eccentric exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate mouth rinsing (Experimental): Rinsing mineral water for 20 seconds
  Interventions: Other: Carbohydrate mouth rinsing
- caffeine gum (Experimental): placebo gum chewing for 10 min
  Interventions: Other: 200 mg caffeine gum

INTERVENTIONS:
Other: Carbohydrate mouth rinsing — the carbohydrate solution was prepared by dissolving 6.4 g of colorless and odorless maltodextrin in 93.6 mL of water; the mixtures were then adjusted to a 6.4% maltodextrin solution for the participants to rinse their mouths for 20 seconds
  Arms: Carbohydrate mouth rinsing
Other: 200 mg caffeine gum — Chewing caffeinated gum for 20 minutes
  Arms: caffeine gum

SUMMARY:
Two experiments were completed to investigate the effects of carbohydrate mouth rinsing and caffeine gum chewing on inertial resistance exercise performance. It was found that both carbohydrate gargling and caffeine gum chewing could improve inertial resistance exercise performance.

DETAILED DESCRIPTION:
This study compared the effects of mouth rinsing with carbohydrates trial (CMR) or a placebo trial (PL) on inertial weight training performance with an inertial weight resistance device. The participants were recruited in this study. Participants were randomly allocated to the CMR and PL groups and subjected to a crossover experiment in which they performed maximum inertial resistance training comprising five sets of six reps, with 3-min rests between sets. After deducting the first repetition of each sets, the mean values from the five sets were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. regular weight training habits,
2. familiarity with Romanian deadlift movements
3. no chronic diseases such as hypertension, diabetes, and kidney disease or sports injuries such as lacerated knee ligaments, inflammation and rupture of tendons, strained biceps femoris or quadriceps, and strained biceps within the 6 months prior.

Exclusion Criteria:

1. did not have regular exercise habits,
2. were unfamiliar with Romanian deadlift movements
3. had certain health problems that prevented them from performing exercise or injury from which they had not recovered for more than 6 months were excluded.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
average power performance of Romanian deadlifts on flywheel training device | immediately after intervention
  average power (watt)
concentric peak power performance of Romanian deadlifts on flywheel training device | immediately after intervention
  concentric peak power (watt)
eccentric peak power performance of Romanian deadlifts on flywheel training device | immediately after intervention
  eccentric peak power (watt)

SECONDARY OUTCOMES:
peak overload performance of Romanian deadlifts on flywheel training device | immediately after intervention
  peak overload (%)
average force performance of Romanian deadlifts on flywheel training device | immediately after intervention
  average force (N)

CONTACTS AND LOCATIONS:
Overall Officials: ChihHui Chiu, PhD, Study Director — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
Only the researcher can see the data

DOCUMENTS (1):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/49/NCT05900349/Prot_000.pdf